CLINICAL TRIAL: NCT03693417
Title: Heated Breathing Circuit on Postoperative Sore Throat After Endobronchial Tube Insertion
Brief Title: Heated Circuit on Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HeatPOSTSingle
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: General Anesthesia
Keywords: pharyngitis; intubation; heat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Device: Heated circuit off
- Heat (Experimental)
  Interventions: Device: Heated circuit on

INTERVENTIONS:
Device: Heated circuit on — Heated circuit will be turned on.
  Arms: Heat
Device: Heated circuit off — Heated circuit will be turned off.
  Arms: Control

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the use of heated breathing circuit in patients undergoing endotracheal intubation for general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for general anesthesia with endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Mallampatti scores greater than 2
* Recent sore throat
* Cervical spine disease
* Recent upper respiratory infection
* Recent analgesics
* History of head and neck surgery
* Friable teeth
* Multiple intubation attempts

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative sore throat for postoperative 24 hour | At 24 hour

SECONDARY OUTCOMES:
Number of participants with postoperative sore throat | At 2, 4, and 24 hour
Number of participants with postoperative hoarseness | At 2, 4, and 24 hour
Wound pain scores | At 2, 4, and 24 hour
  Visual analogue scales will be used (10: most imaginable pain, 0: no pain).

IPD SHARING:
Plan to Share IPD: Undecided